CLINICAL TRIAL: NCT00002269
Title: A Multicenter, Double-Blind, Controlled Study to Evaluate Ampligen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HEM Research (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 073A; AMP-700
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-08

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; ampligen; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — poly(I).poly(c12,U); Zidovudine

INTERVENTIONS:
Drug: Ampligen
Drug: Zidovudine

SUMMARY:
To evaluate ampligen at two dosage levels given twice weekly in combination with zidovudine (AZT) versus AZT alone in individuals with HIV-related immune dysfunction defined as T4 count between 100 and 300 cells/mm3.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositivity.
* Absolute number of T4 cells 100-300 cells/mm3.
* Given informed consent.
* Zidovudine (AZT) therapy for 6 months prior to study entry.
* At least one of the listed HIV-related clinical symptoms or opportunistic infections:
* weight loss > 10 percent, unexplained diarrhea, unexplained intermittent fever, oral candidiasis > 1 month, decreased Karnofsky, oral hairy leukoplakia, chronic fatigue.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Evidence of AIDS.
* Intercurrent acute medical disorder.

Concurrent Medication:

Excluded:

* Chemotherapy for Kaposi's sarcoma (KS).
* Aspirin.
* Non-steroidal anti-inflammatory drugs.

Patients with the following are excluded:

* Inability to return for treatment and evaluation for 12 months.
* Intercurrent acute medical disorder.
* Evidence of AIDS.
* Receiving chemotherapy for Kaposi's sarcoma (KS).
* Unwilling or unable to give informed consent.

Required:

* Zidovudine (AZT).

Required at least 6 months prior to study entry:

* Zidovudine (AZT).

Active drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Oregon Health Sciences Univ, Portland, Oregon
  - MCP Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Nelson Tebedo Community Clinic, Dallas, Texas
  - Dr Patricia Salvato, Houston, Texas